CLINICAL TRIAL: NCT03222583
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of ABT-493/ABT-530 in Treatment-Naïve and Treatment-Experienced, Non-Cirrhotic Asian Adults With Chronic Hepatitis C Virus Genotype (GT) 1 to GT6 Infection With or Without Human Immunodeficiency Virus Co-Infection
Brief Title: A Study to Evaluate the Efficacy and Safety of Glecaprevir/Pibrentasvir (ABT-493/ABT-530) in Treatment-Naive and Treatment-Experienced, Non-Cirrhotic Asian Adults With Chronic Hepatitis C Virus Genotype (GT) 1 to GT6 Infection With or Without Human Immunodeficiency Virus Co-Infection
Acronym: VOYAGE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-592
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C Virus (HCV)
Keywords: Chronic Hepatitis C Virus (HCV); Genotype 1 to 6; Asian; non-cirrhotic; Human Immunodeficiency Virus; co-infection; Treatment-naïve; Treatment-experienced; interferon
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Acquired Immunodeficiency Syndrome; Coinfection | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glecaprevir/Pibrentasvir (Experimental): Participants received oral glecaprevir/pibrentasvir (300 mg/120 mg) once daily with food for 8 or 16 weeks during the double-blind (DB) treatment period.
  Participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
  Interventions: Drug: Glecaprevir/Pibrentasvir
- Placebo / Glecaprevir/Pibrentasvir (Experimental): Participants received placebo to glecaprevir/pibrentasvir for 8 or 16 weeks during the DB treatment period followed by glecaprevir/pibrentasvir (300 mg/120 mg) once daily for 8 or 16 weeks during the open-label (OL) treatment period.
  In each period participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
  Interventions: Drug: Placebo; Drug: Glecaprevir/Pibrentasvir

INTERVENTIONS:
Drug: Placebo — Matching placebo tablet for oral administration
  Arms: Placebo / Glecaprevir/Pibrentasvir
Drug: Glecaprevir/Pibrentasvir — Coformulated tablet for oral administration
  Other Names: ABT-493/ABT-530; MAVYRET™

SUMMARY:
This study will evaluate the efficacy and safety of glecaprevir/pibrentasvir (ABT-493/ABT-530) in non-cirrhotic chronic hepatitis C virus (HCV) genotype (GT)1 to GT6-infected Asian participants with or without human immunodeficiency virus (HIV) co-infection who are HCV treatment-naïve or treatment-experienced with interferon (IFN) with or without ribavirin (RBV), OR sofosbuvir with RBV with or without IFN.

DETAILED DESCRIPTION:
Randomization was stratified by geographic region (China, South Korea, Singapore), genotype (GT1, GT2, combined GT3 - 6), and HCV/HIV co-infection status (co-infected, not co-infected). In China, eligible participants were randomized to Arm A or Arm B (defined below) in the following ratios: 2:1 for GT1, 2:1 for GT2, and 2:1 for combined GT3-6. In South Korea and Singapore, eligible participants were randomized to Arm A or Arm B in the following ratios: 2:1 for GT1 and 2:1 for GT2.

All Primary and Secondary Outcome Measures were pre-specified to be analyzed only in Arm A.

ELIGIBILITY:
Inclusion Criteria:

* Must be of Asian descent
* Screening laboratory result indicating hepatitis C virus (HCV) genotype (GT) 1, 2, 3, 4, 5 or 6 infection.
* Positive anti-HCV antibody (Ab) and HCV ribonucleic acid (RNA) viral load ≥ 1000 IU/ mL at Screening Visit.
* Chronic HCV infection defined as one of the following:

  * Positive for anti-HCV Ab or HCV RNA at least 6 months before Screening; or
  * A liver biopsy consistent with chronic HCV infection
* HCV treatment-naïve to any approved or investigational HCV treatment or treatment-experienced with interferon (IFN) (alpha, beta or pegylated interferon[pegIFN] with or without ribavirin, OR sofosbuvir with RBV with or without IFN. Previous treatment must have been completed ≥ 8 weeks prior to screening.
* Participant must be documented as non-cirrhotic.
* Participants enrolled with human immunodeficiency virus (HIV)-1 and HCV co-infection must also meet the following criteria:

  * Positive test result for human immunodeficiency virus antibody (HIV Ab) at Screening
  * Naïve to treatment with any antiretroviral therapy (ART) with a cluster of differentiation (CD)4+ count greater than or equal to 500 cells/mm³ (or CD4+ percent ≥ 29%)
  * On a stable, qualifying HIV-1 ART regimen with CD4+ count ≥ 200 cells/mm³ (or CD4+ % ≥ 14%) at Screening and plasma HIV-1 RNA below lower limit of quantification (LLOQ) by an approved plasma HIV-1 RNA quantitative assay at Screening and at least once during the 12 months prior to Screening.

Exclusion Criteria:

* Positive test result for Hepatitis B surface antigen (HbsAg) or positive test result for hepatitis B virus (HBV) deoxyribonucleic acid (DNA) if HBsAg is negative.
* Any cause of liver disease other than chronic HCV-infection.
* HCV genotype performed during screening indicating co-infection with more than one HCV genotype
* Clinically significant abnormalities, other than HCV infection or HCV/HIV co-infection
* Chronic human immunodeficiency virus, type 2 (HIV-2) infection

Additional Exclusion Criteria for participants with HCV/HIV Co-Infection:

* For participants on stable ART, taking anti-retroviral agent(s) other than those permitted
* Treatment for an acquired immunodeficiency syndrome (AIDS)-associated opportunistic infection within 12 months of Screening or prophylaxis for an AIDS-associated opportunistic infection within 6 months of screening
* Diagnosis of any clinical AIDS-defining event within 12 months prior to Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (48):
- China (34):
  - Peking University Peoples Hospit /ID# 156846, Beijing, Beijing Municipality
  - Guangzhou Eighth People's Hosp /ID# 156859, Guangzhou, Guangdong
  - Guangdong General Hospital /ID# 156822, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 156860, Guangzhou, Guangdong
  - The Third Affiliated Hospital Of Sun Yat-Sen University /ID# 156900, Guangzhou, Guangdong
  - Xiangya Hospital Central South University /ID# 156901, Changsha, Hunan
  - The Second Hospital of Nanjing /ID# 156863, Nanjing, Jiangsu
  - Jiangsu Province People's Hospital /ID# 156861, Nanjing, Jiangsu
  - The First Hosp of Jilin Univ /ID# 156820, Changchun, Jilin
  - The Sixth People's Hospital of Shenyang /ID# 156849, Shenyang, Liaoning
  - Shanghai Changzheng Hospital /ID# 158072, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong /ID# 157336, Shanghai, Shanghai Municipality
  - Huashan Hospital of Fudan University /ID# 156904, Shanghai, Shanghai Municipality
  - Shanghai Public Health Cli Ctr /ID# 156832, Shanghai, Shanghai Municipality
  - West China Hospital /ID# 156830, Chengdu, Sichuan
  - Beijing Di Tan Hospital, Capital Medical University /ID# 156847, Beijing
  - 1st Hospital of Peking Uni /ID# 156845, Beijing
  - 302 Military Hospital Of China /ID# 156841, Beijing
  - Beijing Friendship Hospital /ID# 156840, Beijing
  - Beijing Youan Hosp, Cap Med Un /ID# 163430, Beijing
  - 1st Affiliated Hosp 3rd Milita /ID# 156831, Chongqing
  - Dalian Sixth Peoples Hospital /ID# 163433, Dalian
  - Mengchao Hepatobiliary Hospita /ID# 156902, Fuzhou
  - Hainan General Hospital /ID# 156839, Haikou, Hainan
  - Jinan Infectious Diseases Hosp /ID# 156886, Jinan, Shandong
  - Chinese People's Liberation Army 81 Hospital /ID# 156862, Nanjing
  - Shengjing Hospital of China Medical University /ID# 156824, Shenyang
  - Tianjin Third Central Hospital /ID# 156816, Tianjin
  - 1st Aff Hosp Xinjiang Med Uni /ID# 156887, Ürümqi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 156884, Wuhan
  - Tongji Hosp Tongji Med College /ID# 156885, Wuhan
  - Fourth Military Medical University Tangdu Hospital, PLA /ID# 156765, Xi'an
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University /ID# 163432, Xi'an
  - Henan Provincial Peoples Hosp /ID# 157197, Zhengzhou, Henan
- Singapore (3):
  - National University Hospital ( /ID# 163272, Singapore
  - Singapore General Hospital /ID# 163271, Singapore
  - Changi General Hospital /ID# 163270, Singapore
- South Korea (11):
  - Pusan National University Hosp /ID# 163371, Busan, Busan Gwang Yeogsi
  - Seoul National Univ Bundang ho /ID# 163367, Seongnam, Gyeonggido
  - Inje University Busan Paik Hospital /ID# 163329, Pusan, Gyeongsangbuk-do
  - Pusan Nat Univ Yangsan Hosp /ID# 163334, Yangsan, Gyeongsangnam-do
  - Inha University Hospital /ID# 163320, Junggu, Incheon Gwang Yeogsi
  - Yonsei University Health System, Severance Hospital /ID# 163339, Seodaemun-gu, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 163364, Seoul, Seoul Teugbyeolsi
  - Cath Univ Seoul St Mary's Hosp /ID# 163341, Seoul, Seoul Teugbyeolsi
  - Korea Universtiy Guro Hospital /ID# 163380, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 163348, Seoul
  - Asan Medical Center /ID# 163336, Seoul

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Wei L, Wang G, Alami NN, Xie W, Heo J, Xie Q, Zhang M, Kim YJ, Lim SG, Fredrick LM, Lu W, Liu W, Kalluri HV, Krishnan P, Tripathi R, Mobashery N, Burroughs M, Asatryan A, Jia J, Hou J. Glecaprevir-pibrentasvir to treat chronic hepatitis C virus infection in Asia: two multicentre, phase 3 studies- a randomised, double-blind study (VOYAGE-1) and an open-label, single-arm study (VOYAGE-2). Lancet Gastroenterol Hepatol. 2020 Sep;5(9):839-849. doi: 10.1016/S2468-1253(20)30086-8. Epub 2020 Jul 16. PMID 32682494

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 47 sites in China, South Korea, and Singapore. Eligible participants were non-cirrhotic chronic hepatitis C (HCV) genotype (GT)1-6-infected adults with or without HIV co-infection who were HCV treatment-naïve or treatment-experienced with regimens containing interferon (IFN), pegylated IFN, ribavirin, and/or sofosbuvir.
Pre-assignment Details: Randomization was stratified by geographic region, genotype (GT1, GT2, combined GT3 - 6), and HCV/HIV co-infection status (co-infected, not co-infected). Participants were randomized to Arm A or Arm B in the following ratios: China: 2:1 for GT1, 2:1 for GT2, and 2:1 for combined GT3 - 6; South Korea and Singapore: 2:1 for GT1 and 2:1 for GT2.
Groups:
- Arm A: Glecaprevir/Pibrentasvir: Participants received oral glecaprevir/pibrentasvir (300 mg/120 mg) once daily with food for 8 or 16 weeks during the double-blind (DB) treatment period.
  Participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
- Arm B: Placebo / Glecaprevir/Pibrentasvir: Participants received placebo to glecaprevir/pibrentasvir for 8 or 16 weeks during the DB treatment period followed by glecaprevir/pibrentasvir (300 mg/120 mg) once daily for 8 or 16 weeks during the open-label (OL) treatment period.
  In each period participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
Period: Overall Study
Arm/Group | Arm A: Glecaprevir/Pibrentasvir | Arm B: Placebo / Glecaprevir/Pibrentasvir
Started | 363 | 183
Received Double-blind Treatment | 362 | 183
Completed Double-blind Period | 360 | 183
Entered Open-label Period (The open-label treatment period was only applicable for participants assigned to Arm B (placebo).) | 0 | 182
Completed Open-label Period | 0 | 181
Completed | 358 | 177
Not Completed | 5 | 6
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug during the DB Treatment Period
Groups:
- Arm A: Glecaprevir/Pibrentasvir: Participants received oral glecaprevir/pibrentasvir (300 mg/120 mg) once daily with food for 8 or 16 weeks during the double-blind (DB) treatment period.
- Arm B: Placebo / Glecaprevir/Pibrentasvir: Participants received placebo to glecaprevir/pibrentasvir for 8 or 16 weeks during the DB treatment period followed by glecaprevir/pibrentasvir (300 mg/120 mg) once daily for 8 or 16 weeks during the open-label (OL) treatment period.
- Total: Total of all reporting groups
Arm/Group | Arm A: Glecaprevir/Pibrentasvir | Arm B: Placebo / Glecaprevir/Pibrentasvir | Total
Number analyzed (Participants) | 362 | 183 | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.68 (12.96) | 49.18 (13.55) | 48.85 (13.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 97 | 277
  Male | 182 | 86 | 268
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 362 | 183 | 545
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 82 | 42 | 124
  Singapore | 21 | 11 | 32
  China | 259 | 130 | 389
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1 | 179 | 89 | 268
  Genotype 2 | 139 | 71 | 210
  Genotype 3 | 26 | 10 | 36
  Genotype 4 | 0 | 1 | 1
  Genotype 5 | 0 | 0 | 0
  Genotype 6 | 18 | 12 | 30
Prior HCV Treatment History [Count of Participants; unit: Participants] — Treatment-experienced includes treatment with interferon (IFN; alpha, beta or pegylated interferon [pegIFN]) with or without ribavirin (RBV), OR sofosbuvir with RBV with or without IFN.
  Participants
    Treatment-naive | 281 | 155 | 436
    Treatment-experienced | 81 | 28 | 109
Human Immunodeficiency Virus (HIV) Co-infection Status [Count of Participants; unit: Participants]
  Hepatitis C infection only | 362 | 183 | 545
  HCV / HIV co-infection | 0 | 0 | 0
HCV Ribonucleic Acid (RNA) Level [Mean (Standard Deviation); unit: log₁₀ IU/mL] | 6.37 (0.72) | 6.26 (0.79) | 6.33 (0.74)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of HCV GT1 - GT6-Infected Participants in Arm A Who Achieved Sustained Virologic Response 12 Weeks Post Treatment (SVR12)
Description: Sustained virologic response 12 weeks post-treatment (SVR12) was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (LLOQ; less than 15 IU/mL) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug, Week 20 or Week 28 depending on the treatment regimen.
Population: This endpoint was pre-specified to be analyzed in participants randomized to Arm A who received at least 1 dose of study drug during the DB Treatment Period. Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backward imputation were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 362
percentage of participants | 97.2
Statistical Analysis 1: Comparison: Arm A: Glecaprevir/Pibrentasvir; In order to control the Type I error rate, a fixed sequence testing procedure was used for the 3 ranked primary efficacy endpoints. Only if success had been demonstrated for the first primary endpoint was testing to proceed to the second primary endpoint. Similarly, only if success had been demonstrated for the second primary endpoint was testing to proceed to the third primary endpoint; Test type: Non-Inferiority — The percentage of participants in Arm A with SVR12 was non-inferior to the historical SVR12 rate of 96% if the lower confidence bound (LCB) of the 2-sided 95% confidence interval (CI) for the percentage was > 90%; Percentage of Participants with SVR12 = 97.2, 95% CI 2-sided [95.5 to 98.9]

2. Primary Outcome: Percentage of HCV GT1-Infected Participants in Arm A Who Achieved SVR12
Description: SVR12 was defined as plasma HCV RNA level less than 15 IU/mL 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after last actual dose of study drug, Week 20 or Week 28 depending on the treatment regimen
Population: This endpoint was pre-specified to be analyzed in GT1-infected participants randomized to Arm A who received at least one dose of study drug. Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backward imputation were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 179
percentage of participants | 99.4
Statistical Analysis 1: Comparison: Arm A: Glecaprevir/Pibrentasvir; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The percentage of GT1-infected participants in Arm A with SVR12 was non-inferior to the historical SVR12 rate of 97% if the LCB of the 2-sided 95% CI for the percentage was > 91%; Percentage of Participants with SVR12 = 99.4, 95% CI 2-sided [98.3 to 100.0]

3. Primary Outcome: Percentage of HCV GT2-Infected Participants in Arm A Who Achieved SVR12
Description: SVR12 was defined as plasma HCV RNA level less than 15 IU/mL 12 weeks after the last actual dose of study drug.
Time Frame: 12 weeks after the last dose of study drug, Week 20 or Week 28 depending on the treatment regimen.
Population: This endpoint was pre-specified to be analyzed in genotype 2-infected participants randomized to Arm A who received at least one dose of study drug. Backward imputation, where applicable, was used to impute missing data. Participants with missing data after backward imputation were counted as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 139
percentage of participants | 97.8
Statistical Analysis 1: Comparison: Arm A: Glecaprevir/Pibrentasvir; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The percentage of GT2-infected participants in Arm A with SVR12 was non-inferior to the historical SVR12 rate of 95% if the LCB of the 2-sided 95% CI for the percentage was > 89%; Percentage of Participants with SVR12 = 97.8, 95% CI 2-sided [95.4 to 100.0]

4. Secondary Outcome: Percentage of Participants in Arm A With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as meeting one of the following:
  * confirmed increase from nadir in HCV RNA (two consecutive HCV RNA measurements > 1 log₁₀ IU/mL above nadir) at any time point during the treatment period; or
  * confirmed HCV RNA greater than or equal to 100 IU/mL after HCV RNA < 15 IU/mL during the treatment period, or
  * HCV RNA ≥ 15 IU/mL at end of treatment with at least 6 weeks of treatment.
Time Frame: 8 or 16 weeks depending on the treatment regimen
Population: This endpoint was pre-specified to be analyzed in all participants randomized to Arm A who received at least 1 dose of study drug during the DB Treatment Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 362
percentage of participants | 0.6 [0.2 to 2.0]

5. Secondary Outcome: Percentage of Participants in Arm A With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA greater than or equal to 15 IU/mL between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < 15 IU/mL at the end of treatment, excluding re-infection.
Time Frame: From the end of treatment (Weeks 8 or 16) through 12 weeks after the last dose of study drug (Weeks 20 or 28 depending on the treatment regimen).
Population: This endpoint was pre-specified to be analyzed in all participants randomized to Arm A who received at least one dose of study drug, with HCV RNA < 15 IU/mL at the end of treatment, at least one post-treatment HCV RNA value, and who completed the assigned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 359
percentage of participants | 1.7 [0.8 to 3.6]

6. Secondary Outcome: Percentage of HCV/HIV Co-infected Participants in Arm A Who Achieved SVR12
Description: SVR12 was defined as plasma HCV RNA level less than 15 IU/mL 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug, Week 20 or 28 depending on the treatment regimen
Population: No HCV-HIV co-infected participants were enrolled in the study
Arm/Group | Arm A: Glecaprevir/Pibrentasvir
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Double-blind Treatment Period: From initiation of study drug through 30 days after last dose and prior to Day 1 of the open-label period, if applicable; up to 12 or 20 weeks depending on the treatment regimen. Open-label Treatment Period (Arm B only): From the first dose of study drug in the OL period up to 30 days after the last dose of OL study drug; up to 12 or 20 weeks depending on the treatment regimen.
Groups:
- DB Period: Arm A - Glecaprevir/Pibrentasvir: Participants received oral glecaprevir/pibrentasvir (300 mg/120 mg) once daily with food for 8 or 16 weeks during the double-blind (DB) treatment period.
  Participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
- DB Period: Arm B - Placebo: Participants received placebo to glecaprevir/pibrentasvir for 8 or 16 weeks during the DB treatment period.
  Participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
- OL Period: Arm B - Glecaprevir/Pibrentasvir: Participants randomized to receive placebo in the DB treatment period received glecaprevir/pibrentasvir (300 mg/120 mg) once daily for 8 or 16 weeks during the open-label (OL) treatment period.
  Participants received treatment for 8 weeks with the exception of treatment-experienced, genotype 3-infected participants who received treatment for 16 weeks.
Arm/Group | DB Period: Arm A - Glecaprevir/Pibrentasvir | DB Period: Arm B - Placebo | OL Period: Arm B - Glecaprevir/Pibrentasvir
All-Cause Mortality (participants affected / at risk) | 0/362 | 0/183 | 0/182
Serious Adverse Events (participants affected / at risk) | 3/362 | 4/183 | 5/182
Other Adverse Events (participants affected / at risk) | 36/362 | 18/183 | 22/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Arm A - Glecaprevir/Pibrentasvir (N=362) | DB Period: Arm B - Placebo (N=183) | OL Period: Arm B - Glecaprevir/Pibrentasvir (N=182)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Arm A - Glecaprevir/Pibrentasvir (N=362) | DB Period: Arm B - Placebo (N=183) | OL Period: Arm B - Glecaprevir/Pibrentasvir (N=182)
Upper respiratory tract infection (Infections and infestations) | 36 (36) | 18 (18) | 22 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03222583/SAP_000.pdf
  • Study Protocol (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT03222583/Prot_001.pdf